CLINICAL TRIAL: NCT04700514
Title: Effect of Anesthetic Drugs on Neurocognitive Function in Children With Retinoblastoma Requiring Multiple Anesthetic Exposure - Preliminary Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Clinical Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2009-039-1155
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 1. Children diagnosed with retinoblastoma and received exam under anesthesia (EUA) before the age of 30 months, and is not yet 4 years old
  2. Children who are undergoing exams and treatment such as EUA, chemoport insertion, or intra-arterial chemotherapy under general anesthesia
  3. Sevoflurane is used only for anesthesia
- Dexmedetomidine group (Experimental): 1. Children who are diagnosed with retinoblastoma and are scheduled for the first EUA before their age of 30 months.
  2. No history of anesthesia
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine (1 mcg/kg loading for 10 min, then 1 mcg/kg/min continuous infusion) is used with sevoflurane in every time of general anesthesia
  Arms: Dexmedetomidine group

SUMMARY:
This study evaluate the effect of dexmedetomidine on intelligence test in pediatric patients with multiple anesthesia exposure. Children who are diagnosed with retinoblastoma and receive first exam under general anesthesia before age of 2 are included. Intelligence test will performed when patients' age are 4.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are first diagnosed as retinoblastoma and scheduled for EUA and treatment under general anesthesia before age of 2

Exclusion Criteria:

-

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
IQ score at age of 4 | year 4
  Korean-Wechsler Preschool and Primary Scale of Intelligence test (score >131, high; score 116-130, high-normal; socre 85-115, normal; score 70-84; low-normal; score <69; low)
Developmental Test | year 4
  visual-Motor Integration test

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea